CLINICAL TRIAL: NCT02169037
Title: Substrate Ablation (Focal Impulse and Rotor Modulation) Compared to Pulmonary Vein Isolation to Eliminate Paroxysmal Atrial Fibrillation: A Randomized Clinical Trial
Brief Title: Substrate Versus Trigger Ablation for Paroxysmal Atrial Fibrillation
Acronym: SUBSTRATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAR083359; R01HL083359 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
Keywords: Rotor; FIRM; Paroxysmal Atrial Fibrillation; Atrial tachyarrhythmia; Ablation; Contact mapping; Clinical trial; Signal processing.
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FIRM ablation (Experimental): These patients will be treated by ablation of patient-specific rotors and focal sources (FIRM) alone.
  Interventions: Procedure: FIRM Ablation
- Conventional AF ablation with PVI (Active Comparator): These patients will treated by conventional AF ablation by pulmonary vein isolation (PVI) alone.
  Interventions: Procedure: Conventional AF ablation with PVI

INTERVENTIONS:
Procedure: FIRM Ablation — Substrate ablation for AF, via ablation of rotors and focal sources alone.
  Arms: FIRM ablation
Procedure: Conventional AF ablation with PVI — Trigger Based Ablation for AF, using Pulmonary Vein Isolation alone.
  Arms: Conventional AF ablation with PVI

SUMMARY:
This is a prospective randomized study to assess the safety and efficacy of FIRM (Focal Impulse and Rotor Modulation)-guided ablation for the treatment of symptomatic atrial fibrillation (AF). The study hypothesis is that the efficacy of AF elimination at 1 year will be higher by ablating patient-specific AF-sustaining rotors and focal sources by Focal Impulse and Rotor Modulation (FIRM) compared to conventional ablation alone (wide-area PV isolation).

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is a standard of care therapy for atrial fibrillation (AF). However, it produces suboptimal results, with a single procedure success of 45-55%, and multiple procedure success rates of 65-75% in recent randomized trials. The rationale of PVI is to eliminate triggers from the Pulmonary veins. An alternative strategy is to eliminate the substrates that sustain AF after it has been triggered, as applied to other arrhythmias. However, the relevance of AF substrates - at least in persistent AF - has been questioned with the recent STAR-AF-II trial, in which ablating at additional lines or complex atrial electrograms (CFAE) did not improve the success of PVI alone (Verma et al., 2015) - although success remained at ~50% for a single procedure. Because of STAR-AF2, the PVI limb in this trial will be PVI alone (wide area circumferential ablation) with no additional lesions.

Focal Impulse and Rotor Modulation (FIRM) is a novel approach to eliminate specific electrical substrates for AF, demonstrated in studies from many laboratories to take the form of localized electrical circuits. These rotors and focal sources lie in patient-specific locations, often away from typical PVI ablation sites and in right atrium, and ablating them has substantially improved the single procedure success rate of PVI in several multi center non-randomized trials (Narayan, J Am Coll Cardiol. 2012; Miller, J Cardiovasc Electrophysiol. 2014).

There is therefore equipoise in the literature between PVI alone, with a long-history but suboptimal results, and FIRM only, that is newer with potentially greater efficacy but without randomized trial data.

This study will test both strategies in a randomized controlled fashion.

ELIGIBILITY:
INCLUSION CRITERIA:

* male or female >21 years
* reported incidence of at least two documented episodes of symptomatic paroxysmal atrial fibrillation (AF) during the three months preceding trial entry (at least 1 episode documented by 12-lead ECG or ECG rhythm strip)
* women without childbearing potential or women of childbearing potential who are not pregnant per a serum HCG test
* refractory to at least one Class I or III anti-arrhythmic medications. Drug doses must be therapeutic and stable
* willingness, ability and commitment to participate in baseline and follow-up evaluations without participation in another clinical trial (unless documented approval received from both sponsors)
* oral anticoagulation required for those subjects who have a score of two or more based on the following criteria (CHAD score):

  * Congestive heart failure (1 point)
  * hypertention (1 point)
  * age 75 years or older (2 points)
  * diabetes (1 point)
  * prior stroke or transient ischemic attack (2 points)
  * vascular disease (1 point)
  * age 65 years or older (1 point)
  * sex category: female (1 point)
* patient is willing and able to remain on anti-coagulation therapy for a minimum of 3 months post procedure for all subjects, and potentially indefinitely post procedure if the patient has CHAD score >or=2
* signed informed consent after a full discussion of the risks and benefits of both therapy arms, and the concept of randomization
* NYHA Class 0,I, II stable on medical therapy for > 3months
* left atrial diameter <or= 5.5cm
* LVEF >or=40%
* sustained AF during the procedure

EXCLUSION CRITERIA:

* atrial fibrillation from a reversible cause (e.g., surgery, hyperthyroidism, pericarditis)
* cardiac or thoracic surgery within the past 180 days
* AF secondary to electrolyte imbalance, thyroid disease
* contraindication to Heparin
* Contraindication to Warfarin or other novel oral anticoagulants
* history of significant bleeding abnormalities
* history of significant blood clotting abnormalities, systemic thrombi or systemic embolization
* ASD closure device, LAA closure device, prosthetic mitral or tricuspid valve
* atrial clot/thrombus on imaging such as on a trans-esophageal echocardiogram (TEE) within 72 hours of the procedure
* intramural thrombus or other cardiac mass that may adversely effect catheter introduction or manipulation
* significant pulmonary embolus within 6 months of enrollment
* acute illness or active systemic infection or sepsis that may ordinarily warrant postponement of the procedure
* history of recent cerebrovascular disease (stroke or TIA) or systemic thromboembolism within < 6 months
* NYHA classes III, IV
* heart failure that is not stable on medical therapy
* pulmonary edema, that may make planned anesthesia or sedation difficult
* stable/unstable angina or ongoing myocardial ischemia
* myocardial infarction (MI) within the past three months
* structural heart disease of clinical significance including:

  * congenital heart disease where the abnormality or its correction prohibit or increase the risk of ablation
  * acquired heart disease that may increase risk of ablation, such as significant ventricular septal defect post myocardial infarction
  * rheumatic valve disease, since this produces a unique AF phenotype
  * extreme left atrial enlargement (LA volume index > 60 ml/m2) in whom PVI has low success and 55 mm baskets are too small for the atria
* cardiac transplantation or other cardiac surgery planned within the 12 month followup period of the trial
* life expectancy less than 12 months (the followup period of the trial)
* significant pulmonary disease (e.g., COPD) or any other disease that significantly increase the risk to the patient from sedation or anesthesia
* untreatable allergy to contrast media
* at time of ablation procedure, clinically significant abnormalities in serum potassium, sodium, magnesium or other electrolytes that affect the suitability of the patient for ablation at that time

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Long term success | 12 months
  Freedom from AF recurrence during 12 months after the initial AF ablation procedure, after an initial 3 month blanking (healing and stabilization) period

SECONDARY OUTCOMES:
Long-term freedom from AF/AT | 12 months
  Freedom from AF and atrial tachycardia (AT) during 12 months after the initial AF ablation procedure, after an initial 3 month blanking (healing and stabilization) period. Atrial tachycardias (AT) include those arising from atrial regions where ablation was performed (such as left atrial tachycardia) as well as from regions where ablation was not performed (such as typical cavotricuspid isthmus dependent atrial flutter).
Total ablation time | 1 day
  Time from first ablation lesion to the last lesion. Total ablation time will be recorded in all patients, measured as the cumulative application of energy from the first ablation lesion to the last lesion. These values will be compared between the FIRM-guided and conventional ablation groups. If ablation for AT/atrial flutter is pursued, this ablation time will be documented separately.
Quality of life (QOL) | 12 months
  Quantitative EuroQol EQ5D scores post-ablation will be compared to those pre-ablation at all time points separately and together (ANOVA).
Adverse events | 12 months
  Adverse events will be adjudicated by an independent Data and Safety Monitoring Board, who will determine whether they are or are not related to the procedure. The number and type of adverse events will be compared between FIRM-guided and conventional ablation groups.
Consistency of Sources At Repeat Ablation | 2 years
  Any patient with a recurrence who consents to restudy will have an assessment of whether rotors and focal sources lie at the same locations as they did at original study.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv M Narayan, MD, PhD, Study Director — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - VA San Diego Medical Center, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883
- [Background] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Background] Narayan SM, Baykaner T, Clopton P, Schricker A, Lalani GG, Krummen DE, Shivkumar K, Miller JM. Ablation of rotor and focal sources reduces late recurrence of atrial fibrillation compared with trigger ablation alone: extended follow-up of the CONFIRM trial (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation). J Am Coll Cardiol. 2014 May 6;63(17):1761-8. doi: 10.1016/j.jacc.2014.02.543. Epub 2014 Mar 13. PMID 24632280
- [Background] Miller, J. M., R. C. Kowal, V. Swarup, J. P. Daubert, E. G. Daoud, J. D. Day, K. A. Ellenbogen, J. D. Hummel, T. Baykaner, D. E. Krummen, S. M. Narayan, V. Y. Reddy, K. Shivkumar, J. S. Steinberg and K. R. Wheelan (2014).